CLINICAL TRIAL: NCT00720434
Title: A Phase 2, Randomized, Placebo Controlled, Dose Ranging Study To Evaluate Peginterferon Alfa 2a (Pegasys®) And Ribavirin (Copegus®) With And Without PF-00868554 In Subjects Chronically Infected With Hepatitis C Virus
Brief Title: A Dose Ranging Study Of PF-00868554 In Combination With PEGASYS And COPEGUS In Patients With Chronic Hepatitis C Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8121007
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — filibuvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): 500 mg BID
  Interventions: Drug: PF-00868554
- B (Experimental): 300 mg BID
  Interventions: Drug: PF-00868554
- C (Experimental): 200 mg BID
  Interventions: Drug: PF-00868554
- D (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-00868554 — 500 mg BID administered as 5x100 mg tablets for 4 weeks in combination with standard of care; standard of care continued for an additional 44 weeks.
  Arms: A
Drug: PF-00868554 — 300 mg BID administered as 3x100 mg tablets for 4 weeks in combination with standard of care; standard of care continued for an additional 44 weeks
  Arms: B
Drug: PF-00868554 — 200 mg BID administered as 2x100 mg tablets for 4 weeks in combination with standard of care; standard of care continued for an additional 44 weeks
  Arms: C
Drug: Placebo — Placebo administered for 4 weeks in combination with standard of care; standard of care continued for an additional 44 weeks
  Arms: D

SUMMARY:
The purpose of this study is to further assess the potency of PF-00868554, an HCV polymerase inhibitor, in subjects chronically infected with HCV by evaluating the antiviral activity of PF-00868554 in combination with current standard of care therapy, pegylated interferon-alpha2a (PEGASYS) and ribavirin (COPEGUS).

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive (no prior treatment with IFN-a +/- RBV regimens.
* Subjects who have discontinued IFN-a containing regimens after <2 weeks of therapy due to tolerability issues are considered treatment naive.
* HCV RNA > 100,000 IU/mL at screening.
* Genotype 1.
* A diagnosis of chronic HCV infection for at least 6 months.

Exclusion Criteria:

* Evidence of acute or chronic infection with HIV or HBV.
* Exposure within the previous three months to an investigational anti-HCV agent.
* Evidence of severe or decompensated liver disease.
* Subjects with liver disease unrelated to HCV infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (8):
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
- Pfizer Investigational Site, Santurce, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121007&StudyName=A%20Dose%20Ranging%20Study%20Of%20PF-00868554%20In%20Combination%20With%20PEGASYS%20And%20COPEGUS%20In%20Patients%20With%20Chronic%20Hepatitis%20C%20Genotype%201%20Infection

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00868554 200 mg + pegIFN Alfa-2a/RBV: PF-00868554 200 milligram (mg) (2 PF-00868554 100 mg tablets) orally twice daily in combination with standard of care during Week 1 to 4 in blinded treatment period, followed by standard of care as per investigator's discretion up to Week 48, then off-treatment up to Week 72 in open-label period. Standard of care included pegylated interferon alfa-2a (pegIFN alfa-2a) 180 microgram (mcg) subcutaneously once weekly starting from Day 1 and ribavirin (RBV) 1000 mg/day tablet orally in 2 divided doses for participants weighing less than or equal to (<=) 75 kilogram (kg); 1200 mg/day orally in 2 divided doses for participants weighing greater than (>) 75 kg.
- PF-00868554 300 mg + pegIFN Alfa-2a/RBV: PF-00868554 300 mg (3 PF-00868554 100 mg tablets) orally twice daily in combination with standard of care during Week 1 to 4 in blinded treatment period, followed by standard of care as per investigator's discretion up to Week 48, then off-treatment up to Week 72 in open-label period. Standard of care included pegIFN alfa-2a 180 mcg subcutaneously once weekly starting from Day 1 and RBV 1000 mg/day tablet orally in 2 divided doses for participants weighing <=75 kg; 1200 mg/day orally in 2 divided doses for participants weighing >75 kg.
- PF-00868554 500 mg + pegIFN Alfa-2a/RBV: PF-00868554 500 mg (5 PF-00868554 100 mg tablets) orally twice daily in combination with standard of care during Week 1 to 4 in blinded treatment period, followed by standard of care as per investigator's discretion up to Week 48, then off-treatment up to Week 72 in open-label period. Standard of care included pegIFN alfa-2a 180 mcg subcutaneously once weekly starting from Day 1 and RBV 1000 mg/day tablet orally in 2 divided doses for participants weighing <=75 kg; 1200 mg/day orally in 2 divided doses for participants weighing >75 kg.
- Placebo + pegIFN Alfa-2a/RBV: Placebo matched to PF-00868554 tablets orally twice daily in combination with standard of care during Week 1 to 4 in blinded treatment period, followed by standard of care as per investigator's discretion up to Week 48, then off-treatment up to Week 72 in open-label period. Standard of care included pegIFN alfa-2a 180 mcg subcutaneously once weekly starting from Day 1 and RBV 1000 mg/day tablet orally in 2 divided doses for participants weighing <=75 kg; 1200 mg/day orally in 2 divided doses for participants weighing >75 kg.
Period: Double-Blind Period (Week 1-4)
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV
Started | 10 | 9 | 8 | 8
Completed | 10 | 8 | 8 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Open-Label Period (Week 5-72)
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV
Started | 10 | 8 | 8 | 8
Completed | 4 | 5 | 4 | 4
Not Completed | 6 | 3 | 4 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Other | 4 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV | Total
Number analyzed (Participants) | 10 | 9 | 8 | 8 | 35
Age, Customized [Number; unit: participants]
  18 to 44 years | 5 | 3 | 3 | 1 | 12
  45 to 64 years | 5 | 6 | 5 | 7 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 2 | 5 | 17
  Male | 7 | 2 | 6 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 4 - Full Analysis Set
Description: Plasma HCV RNA levels were measured using the Roche COBAS Taqman assay (limit of detection: 25 international unit per milliliter [IU/mL]). Baseline value calculated as the average of the screening and Day 1 pre-dose measurements.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug and had both baseline and at least 1 valid post-baseline endpoint measurements for HCV viral load. Here 'n' signifies participants evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV
Number analyzed (Participants) | 10 | 9 | 8 | 8
log10 IU/mL
  Baseline (n=10, 9, 8, 8) | 6.38843 (0.483283) | 6.67823 (0.472198) | 6.66254 (0.563548) | 6.42047 (0.499677)
  Change at Week 4 (n=10, 8, 8, 8) | -4.45887 (1.422134) | -4.64646 (1.982243) | -3.61918 (2.488935) | -2.10239 (1.429056)
Statistical Analysis 1: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; An analysis of covariance (ANCOVA) model was used to compare differences among treatments. Independent variables included treatment and log-transformed baseline HCV viral load. Adjusted mean difference and corresponding 95 percentage (%) confidence interval (CI) were calculated; Test type: Superiority or Other; p = 0.0131, ANCOVA; Adjusted Mean Difference = -2.36357, 95% CI 2-sided [-4.19228 to -0.53485]
Statistical Analysis 2: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; An ANCOVA model was used to compare differences among treatments. Independent variables included treatment and log-transformed baseline HCV viral load. Adjusted mean difference and corresponding 95% CI were calculated; Test type: Superiority or Other; p = 0.0142, ANCOVA; Adjusted Mean Difference = -2.49190, 95% CI 2-sided [-4.44619 to -0.53760]
Statistical Analysis 3: Comparison: PF-00868554 500 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1368, ANCOVA; Adjusted Mean Difference = -1.46325, 95% CI 2-sided [-3.41898 to 0.49248]
Statistical Analysis 4: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3321, ANCOVA; Adjusted Mean Difference = -0.90032, 95% CI 2-sided [-2.76711 to 0.96648]
Statistical Analysis 5: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2839, ANCOVA; Adjusted Mean Difference = -1.02865, 95% CI 2-sided [-2.95573 to 0.89844]
Statistical Analysis 6: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 300 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8891, ANCOVA; Adjusted Mean Difference = 0.12833, 95% CI 2-sided [-1.73676 to 1.99342]

2. Secondary Outcome: Proportion of Participants Achieving Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: Proportion of participants achieving undetectable plasma HCV RNA at Week 4 (rapid virologic response), at Week 12 (early virologic response), at Week 48 (end of treatment response), at Week 60 (sustained virologic response; 12 weeks after cessation of therapy), at Week 72 (sustained virologic response; 24 weeks after cessation of therapy) were summarized. Undetectable viral load was defined as HCV RNA <25 IU/mL.
Time Frame: Week 4, 12, 48, 60, 72
Population: Modified Analysis Set: subset of FAS that included all participants who completed the Week 4 visit.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV
Number analyzed (Participants) | 10 | 8 | 8 | 8
proportion of participants
  Week 4 | 0.6000 [0.2624 to 0.8784] | 0.7500 [0.3491 to 0.9681] | 0.6250 [0.2449 to 0.9148] | 0.0000 [0.0000 to 0.3694]
  Week 12 | 0.8000 [0.4439 to 0.9748] | 0.8750 [0.4735 to 0.9968] | 0.6250 [0.2449 to 0.9148] | 0.5000 [0.1570 to 0.8430]
  Week 48 | 0.6000 [0.2624 to 0.8784] | 0.7500 [0.3491 to 0.9681] | 0.6250 [0.2449 to 0.9148] | 0.5000 [0.1570 to 0.8430]
  Week 60 | 0.3000 [0.0667 to 0.6525] | 0.5000 [0.1570 to 0.8430] | 0.5000 [0.1570 to 0.8430] | 0.5000 [0.1570 to 0.8430]
  Week 72 | 0.3000 [0.0667 to 0.6525] | 0.5000 [0.1570 to 0.8430] | 0.5000 [0.1570 to 0.8430] | 0.5000 [0.1570 to 0.8430]
Statistical Analysis 1: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; Week 4: The difference in proportions between treatment groups presented along with 95% CI, were based on exact method for small samples from the binomial distribution; Test type: Superiority or Other; Difference in Proportions = 0.6000, 95% CI 2-sided [0.1565 to 0.8785]
Statistical Analysis 2: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Proportions = 0.7500, 95% CI 2-sided [0.2330 to 0.9690]
Statistical Analysis 3: Comparison: PF-00868554 500 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Proportions = 0.6250, 95% CI 2-sided [0.0871 to 0.9191]
Statistical Analysis 4: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Proportions = -0.0250, 95% CI 2-sided [-0.4769 to 0.4336]
Statistical Analysis 5: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Proportions = 0.1250, 95% CI [-0.4024 to 0.6049]
Statistical Analysis 6: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 300 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Proportions = -0.1500, 95% CI 2-sided [-0.5729 to 0.3149]
Statistical Analysis 7: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; Week 12: The difference in proportions between treatment groups presented along with 95% CI, were based on exact method for small samples from the binomial distribution; Test type: Superiority or Other; Difference in Proportions = 0.3000, 95% CI 2-sided [-0.1836 to 0.6931]
Statistical Analysis 8: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Difference in Proportions = 0.3750, 95% CI 2-sided [-0.1732 to 0.7797]
Statistical Analysis 9: Comparison: PF-00868554 500 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Difference in Proportions = 0.1250, 95% CI 2-sided [-0.4024 to 0.6049]
Statistical Analysis 10: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Difference in Proportions = 0.1750, 95% CI 2-sided [-0.2934 to 0.5917]
Statistical Analysis 11: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Difference in Proportions = 0.2500, 95% CI 2-sided [-0.2913 to 0.6960]
Statistical Analysis 12: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 300 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; Difference in Proportions = -0.0750, 95% CI 2-sided [-0.5144 to 0.3880]
Statistical Analysis 13: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; Week 48: The difference in proportions between treatment groups presented along with 95% CI, were based on exact method for small samples from the binomial distribution; Test type: Superiority or Other; Difference in Proportions = 0.1000, 95% CI 2-sided [-0.3728 to 0.5414]
Statistical Analysis 14: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Difference in Proportions = 0.2500, 95% CI 2-sided [-0.2913 to 0.6960]
Statistical Analysis 15: Comparison: PF-00868554 500 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Difference in Proportions = 0.1250, 95% CI 2-sided [-0.4024 to 0.6049]
Statistical Analysis 16: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Difference in Proportions = -0.0250, 95% CI [-0.4769 to 0.4336]
Statistical Analysis 17: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Difference in Proportions = 0.1250, 95% CI 2-sided [-0.4024 to 0.6049]
Statistical Analysis 18: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 300 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; Difference in Proportions = -0.1500, 95% CI 2-sided [-0.5729 to 0.3149]
Statistical Analysis 19: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; Week 60: The difference in proportions between treatment groups presented along with 95% CI, were based on exact method for small samples from the binomial distribution; Test type: Superiority or Other; Difference in Proportions = -0.2000, 95% CI 2-sided [-0.6191 to 0.2811]
Statistical Analysis 20: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; Difference in Proportions = 0.0000, 95% CI 2-sided [-0.5070 to 0.5070]
Statistical Analysis 21: Comparison: PF-00868554 500 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; Difference in Proportions = 0.0000, 95% CI 2-sided [-0.5070 to 0.5070]
Statistical Analysis 22: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; Difference in Proportions = -0.2000, 95% CI 2-sided [-0.6191 to 0.2811]
Statistical Analysis 23: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; Difference in Proportions = 0.0000, 95% CI 2-sided [-0.5070 to 0.5070]
Statistical Analysis 24: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 300 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; Difference in Proportions = -0.2000, 95% CI 2-sided [-0.6191 to 0.2811]
Statistical Analysis 25: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; Week 72: The difference in proportions between treatment groups presented along with 95% CI, were based on exact method for small samples from the binomial distribution; Test type: Superiority or Other; Difference in Proportions = -0.2000, 95% CI 2-sided [-0.6191 to 0.2811]
Statistical Analysis 26: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; Difference in Proportions = 0.0000, 95% CI 2-sided [-0.5070 to 0.5070]
Statistical Analysis 27: Comparison: PF-00868554 500 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; Difference in Proportions = 0.0000, 95% CI 2-sided [-0.5070 to 0.5070]
Statistical Analysis 28: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; Difference in Proportions = -0.2000, 95% CI 2-sided [-0.6191 to 0.2811]
Statistical Analysis 29: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; Difference in Proportions = 0.0000, 95% CI 2-sided [-0.5070 to 0.5070]
Statistical Analysis 30: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 300 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; Difference in Proportions = -0.2000, 95% CI 2-sided [-0.6191 to 0.2811]

3. Secondary Outcome: Alanine Aminotransferase (ALT) Levels
Time Frame: Week 4, 12, 48, 72
Population: FAS included all randomized participants who received at least 1 dose of study drug and had both baseline and at least 1 valid post-baseline endpoint measurements for HCV viral load. Here 'n' signifies participants evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV
Number analyzed (Participants) | 10 | 9 | 8 | 8
IU/L
  Week 4 (n=10, 8, 8, 8) | 31.1 (12.74) | 28.5 (13.60) | 51.6 (19.45) | 47.1 (27.68)
  Week 12 (n=10, 7, 8, 8) | 32.9 (15.26) | 29.4 (11.12) | 42.5 (15.09) | 35.6 (19.10)
  Week 48 (n=6, 6, 5, 4) | 35.2 (30.80) | 25.7 (12.61) | 24.4 (19.26) | 148.8 (248.26)
  Week 72 (n=6, 5, 5, 4) | 46.0 (40.54) | 34.0 (27.90) | 21.8 (14.20) | 21.5 (12.77)

4. Secondary Outcome: Population Pharmacokinetics (PK) of PF-00868554
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: 1, 2 and 6 hours post-dose on Day 1; 0 hour (pre-dose) on Day 7, 14, 21; 0 hour (pre-dose), 2, 6 hours post-dose on Day 28
Reporting Status: Not Posted

5. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 4 - Modified Analysis Set
Description: Plasma HCV RNA levels were measured using the Roche COBAS Taqman assay (limit of detection: 25 IU/mL). Baseline value calculated as the average of the screening and Day 1 pre-dose measurements.
Time Frame: Baseline, Week 4
Population: Modified Analysis Set: subset of FAS that included all participants who completed the Week 4 visit.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV
Number analyzed (Participants) | 10 | 8 | 8 | 8
log10 IU/mL | -4.45887 (1.422134) | -4.64646 (1.982243) | -3.61918 (2.488935) | -2.10239 (1.429056)
Statistical Analysis 1: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0131, ANCOVA; Adjusted Mean Difference = -2.36357, 95% CI 2-sided [-4.19228 to -0.53485]
Statistical Analysis 2: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0142, ANCOVA; Adjusted Mean Difference = -2.49190, 95% CI 2-sided [-4.44619 to -0.53760]
Statistical Analysis 3: Comparison: PF-00868554 500 mg + pegIFN Alfa-2a/RBV vs Placebo + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1368, ANCOVA; Adjusted Mean Difference = -1.46325, 95% CI 2-sided [-3.41898 to 0.49248]
Statistical Analysis 4: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3321, ANCOVA; Adjusted Mean Difference = -0.90032, 95% CI 2-sided [-2.76711 to 0.96648]
Statistical Analysis 5: Comparison: PF-00868554 300 mg + pegIFN Alfa-2a/RBV vs PF-00868554 500 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2839, ANCOVA; Adjusted Mean Difference = -1.02865, 95% CI 2-sided [-2.95573 to 0.89844]
Statistical Analysis 6: Comparison: PF-00868554 200 mg + pegIFN Alfa-2a/RBV vs PF-00868554 300 mg + pegIFN Alfa-2a/RBV; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8891, ANCOVA; Adjusted Mean Difference = 0.12833, 95% CI 2-sided [-1.73676 to 1.99342]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-00868554 200 mg + pegIFN Alfa-2a/RBV | PF-00868554 300 mg + pegIFN Alfa-2a/RBV | PF-00868554 500 mg + pegIFN Alfa-2a/RBV | Placebo + pegIFN Alfa-2a/RBV
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/9 | 1/8 | 2/8
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00868554 200 mg + pegIFN Alfa-2a/RBV (N=10) | PF-00868554 300 mg + pegIFN Alfa-2a/RBV (N=9) | PF-00868554 500 mg + pegIFN Alfa-2a/RBV (N=8) | Placebo + pegIFN Alfa-2a/RBV (N=8)
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00868554 200 mg + pegIFN Alfa-2a/RBV (N=10) | PF-00868554 300 mg + pegIFN Alfa-2a/RBV (N=9) | PF-00868554 500 mg + pegIFN Alfa-2a/RBV (N=8) | Placebo + pegIFN Alfa-2a/RBV (N=8)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 4 | 4
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 2 | 1 | 1
Cyst (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 4 | 4 | 5 | 5
Influenza like illness (General disorders) | 0 | 2 | 1 | 2
Injection site erythema (General disorders) | 0 | 2 | 1 | 1
Injection site pruritus (General disorders) | 0 | 1 | 0 | 1
Irritability (General disorders) | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 1 | 2
Product taste abnormal (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Vestibulitis (General disorders) | 0 | 0 | 1 | 0
Alveolar osteitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Areflexia (Nervous system disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0
Headache (Nervous system disorders) | 4 | 6 | 4 | 2
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 2 | 3
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 1 | 4 | 2
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Spermatocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.